CLINICAL TRIAL: NCT03454672
Title: A Prospective, Randomized, Double Arm, Controlled Study With Blinded Assessment to Evaluate the Safety and Effectiveness of the Tixel Fractional System in the Treatment of Periorbital Wrinkles in Comparison With Fractional Laser
Brief Title: A Safety and Effectiveness Study of the Tixel Device, (Fractional Peri-orbital Wrinkles Treatment ) Compared With Laser
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Delay in recruitment as per last protocol amendment due to Covid-19
Sponsor: Novoxel Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLN-0460
Record Dates: First submitted 2018-02-17; First posted 2018-03-06 (Actual); Results first posted 2024-06-20 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Wrinkle
Keywords: periorbital; wrinkles; double-arm; Tixel; Laser; controlled; randomized; double; arm; fractional; resurfacing
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Intervention Model Description: The subjects will be randomly allocated to two equally sized groups, one shall be treated by the Tixel, and the other shall be treated by the laser comparator.
Who Masked: Outcomes Assessor
Masking Description: The assessor shall be blinded to the type of intervention when assessing the outcome of the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Tixel (Experimental): Tixel Treatment.
  Interventions: Device: Tixel
- Laser (Active Comparator): Laser Treatment.
  Interventions: Device: Laser

INTERVENTIONS:
Device: Tixel — Tixel treatment. Between 3-5 treatment sessions according to investigator's review of subject response.
  Other Names: Fractional
  Arms: Tixel
Device: Laser — Tixel treatment. Between 3-5 treatment sessions according to investigator's review of subject response.
  Other Names: Fractional
  Arms: Laser

SUMMARY:
This study is designed to explore the safety and the effectiveness of the Tixel device. This device performs fractional treatment of the skin by applying thermal (heat) energy to the skin. The study shall compare the safety and the effectiveness of the Tixel with the safety and the effectiveness of a laser device which is currently cleared for marketing in the US.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 40-70 years old diagnosed with clinically evident fine (mild) to moderate depth periorbital wrinkling
2. Willingness and ability to comply with all required study activities and protocol requirements.
3. The subject is able to provide written informed consent and perform the study's activities according to HIPAA guidelines and/or Israeli law, depending on each specific study site.

   ___________________________________________________________

Exclusion Criteria:

1. The subject may not undergo treatment by the Tixel or comparator device according to the device's contra-indications for use, as defined in the User Manual and in the Instructions for Use and by any other labeling of the device.
2. Female subjects who are pregnant, or planning to become pregnant, or have given birth less than 3 months ago or are lactating.
3. Subjects with significant exposure to critical amounts of ultraviolet light (Sun tan).
4. Subjects who have had the following treatments:

   1. a prior cosmetic procedure to improve facial rhytides (i.e., rhytidectomy, periorbital or eyelid/eyebrow surgery, brow lift, CO2/Erbium/similar laser/fractional resurfacing, radiofrequency treatment) within 12 months
   2. prior facial treatments with laser, surgical, chemical or light based facial treatments within the previous 6 months, such as for botulinum toxin injections, retinoid, microdermabrasion or prescription level glycolic acid treatments
   3. Injectable filler in area to be treated within 9 months of investigation.
   4. permanent facial implant
5. Any subject who have visible scars that may affect evaluation of response and/or quality of photography.
6. Subjects with any type of active cut, wound, inflammation, lesion (benign, premalignant or malignant) or active bacterial, viral, fungal, or herpetic infection on the skin on the designated treatment sites or in close proximity to it.
7. Existing or history of the following (when discussing skin conditions, refers only to the periorbital sites):

   1. skin malignancy, or any diagnosis of suspected malignancy
   2. Collagen or vascular or bleeding disease
   3. Immunosuppression or autoimmune disease
   4. Erythema with or without blistering
   5. History of post inflammatory hyperpigmentation.
   6. Active Acne Vulgaris, Herpes Simplex Virus (HSV-1), or any existing skin condition/disease that in the investigator's opinion would interfere with the evaluation of the safety of the study treatment.
   7. Any skin pathology which can induce bullous lesions, urticaria, or demonstrate a Koebner phenomenon (psoriasis, lichen planus, etc.).
   8. Any disease that inhibits pain sensation
   9. History of keloid formation, or hypertrophic scarring
   10. Conditions affecting healing rate (i.e. diabetes mellitus I or II, vascular condition, etc.)
   11. neuromuscular disorders
8. Subjects who have used, within 30 days, any medication that can cause dermal hypersensitivity or affect skin characteristics (i.e. topically applied Retinoids, Hydroquinone, Chemical peel of any strength: glycolic acid, lactic acid, salicylic acid)
9. Subjects who have used, systemic treatment which may induce dyspigmentation, such as amiodarone, clofazinmine, minocycline or chloroquine.
10. Subjects currently taking or have taken an oral retinoid in the past six months (risk of scarring with therapy); Subjects currently taking long-term oral steroid treatment (causing fragility of the skin, risk of hematoma and bullae formation); Subjects taking Isotretinoin (Accutane or Roaccutan) within past 12 months.
11. Concurrent therapy that, in the principal investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study treatment.
12. Subjects who anticipate the need for surgery or overnight hospitalization during the study.
13. Enrollment in any active study involving the use of investigational devices or drugs.
14. Any other cause per the principal investigator's discretion.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arielle NB Kauvar, M.D, Principal Investigator — New York Laser & Skin Care Clinic; Sharon Naim, B.Sc,, Study Director — Novoxel Ltd.; Rafi Carasso, M.D, Principal Investigator — Hillel Yaffe Medical Center
Locations (2):
- New York Laser & Skin Care, New York, New York, United States
- Dr. Artzi Skin Center Clinic - Linked to Hillel Yaffe Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Laser: Laser Treatment.
  Laser: Laser treatment. Between 3-5 treatment sessions according to investigator's review of subject response.
Period: Overall Study
Arm/Group | Tixel | Laser
Started | 34 | 34
Completed | 25 | 22
Not Completed | 9 | 12
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 1 | 3
Not completed — painful | 1 | 2
Not completed — Non-compliance | 2 | 4
Not completed — personal reasons | 3 | 2
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: 68 subjects were enrolled. They were randomly split into two arms (34/arm) in each site and underwent periorbital fractional treatments.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tixel | Laser | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 31 | 63
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.44 (7.16) | 53.79 (7.29) | 54.11 (7.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 30 | 64
  Male | 0 | 4 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 32 | 30 | 62
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34
  Israel | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Mean Change by Blinded Assessor Evaluation by Fitzpatrick Classification of Facial Wrinkling (FWCS) Scale
Description: The FWCS shall be assessed and quantified by 3 blinded assessors comparing baseline visit to +42 weeks visit.
Time Frame: baseline, 42 Weeks
Population: The images have been presented to the blinded assessors in pairs, in which the treatment arm allocation was masked.
Measure: Mean (Standard Deviation); unit: FWCS units on scale
Arm/Group | Tixel | Laser
Number analyzed (Participants) | 24 | 22
FWCS units on scale | 1.6 (0.6) | 1.7 (0.8)

2. Secondary Outcome: Mean Change of Subject Experience as Measured by Subject's Subjective Satisfaction Score
Description: Subjective satisfaction is scored on a scale from 1-5, from excellent (5-very satisfied) to poor (1-poor or not satisfied at all). compring results from baseline to 42 weeks.
  total minimum total score - 3, total maximum score - 15
Time Frame: Treatment 1 (Baseline), Treatment 4 (Week 12), Treatment 5 (Week 16), Follow-up Visit 1 (Week 20), Follow-up Visit 3 (Week 42)
Population: Each patient's subjective opinion regarding the overall satisfaction with treatment, was measured every visit. The measurement scale contained 5-points: from excellent (5-very satisfied) to poor (1-poor or not satisfied at all). The calculated total score of the 3 questions ("improvement", "treatment experience", "expectations") is presented. the minimum score can be - 3, and the maximum score can be - 15
Measure: Mean (Standard Deviation); unit: Total Calculated Score on a Scale
Arm/Group | Tixel | Laser
Number analyzed (Participants) | 25 | 22
Total Calculated Score on a Scale
  total score Treatment 1 | 9.4 (3.5) | 9.1 (3.2)
  total score Treatment 4 | 11.4 (2.9) | 10.1 (3.1)
  total score Treatment 5 | 11.7 (3.0) | 10.7 (3.5)
  total score FU1 month | 11.4 (3.3) | 11.0 (3.2)
  total score FU3 months | 11.8 (2.5) | 10.8 (3.3)

3. Secondary Outcome: Number of Days Reported by Subject Using Subjective Subject Downtime Assessment
Description: This assessment determines the number of days required for the subject to return to normal, daily activities. This will be assessed at each treatment visit : visit 1 - visit 5.
  The downtime assessment was evaluated after each Tixel treatment visit. The therapist asked the subject in the next visit regarding the 3 parameters that relate to the total downtime assessment.
  The parameters were:
  1. Return to work (Days)
  2. Return to social activities (Days)
  3. Scabs (Days)
  The results for subjective Downtime assessments were grouped by two categories:
  * More than 2 days vs. less or equal to 2 days for Return to work, Return to social activities, Redness, Edema, and Scabs.
  * More than 4 hours vs. less or equal to 4 hours for sensation of heat.
Time Frame: visit 1 - visit 5
Population: Chi-square test was applied to show if the difference of distribution between treatment groups.
Measure: Number; unit: participants
Arm/Group | Tixel | Laser
Number analyzed (Participants) | 24 | 22
participants
  Treatment 1 -Return to work - more that 2 days | 5 | 4
  Treatment 1 - Return to social activities more than 2 days | 7 | 7
  Treatment 1- Redness- more than 2 days | 14 | 13
  Treatment 1- Edema- more than 2 days | 12 | 9
  Tretatment 1 - Scabs - More than 2 days | 17 | 6
  Treatment 1- Sensation of heat- more than 4 hours | 2 | 6
  Treatment 2 -Return to work - more that 2 days | 3 | 4
  Treatment 2 - Return to social activities more than 2 days | 4 | 5
  Treatment 2- Redness- more than 2 days | 12 | 12
  Treatment 2- Edema- more than 2 days | 10 | 6
  Treatment 2- Scabs- more than 2 days | 16 | 6
  Treatment 2- Sensation of heat- more than 4 hours | 0 | 1
  Treatment 3 -Return to work - more that 2 days | 4 | 5
  Treatment 3 - Return to social activities more than 2 days | 4 | 5
  Treatment 3- Redness- more than 2 days | 8 | 8
  Treatment 3- Edema- more than 2 days | 8 | 8
  Treatment 3- Scabs- more than 2 days | 9 | 3
  Treatment 3- Sensation of heat- more than 4 hours | 1 | 3
  Treatment 4 -Return to work - more that 2 days | 4 | 6
  Treatment 4 - Return to social activities more than 2 days | 4 | 6
  Treatment 4- Redness- more than 2 days | 9 | 10
  Treatment 4- Edema- more than 2 days | 9 | 7
  Treatment 4- Scabs- more than 2 days | 10 | 2
  Treatment 4- Sensation of heat- more than 4 hours | 1 | 2
  Treatment 5 -Return to work - more that 2 days | 4 | 2
  Treatment 5 - Return to social activities more than 2 days | 6 | 3
  Treatment 5- Redness- more than 2 days | 10 | 5
  Treatment 5- Edema- more than 2 days | 9 | 6
  Treatment 5- Scabs- more than 2 days | 9 | 1
  Treatment 5- Sensation of heat- more than 4 hours | 0 | 1

4. Secondary Outcome: Pain Level as Measured by the Visual Analog Scale (VAS) Scale
Description: Secondary Safety- VAS is scored on a scale from 0-10, with 0 indicating no pain and 10 indicating worst pain. This will be assessed at each treatment over 8 weeks to 16 weeks (Depending on number of Treatments given).
Time Frame: treatment 1 - treatment 5
Population: The pain level was evaluated immediately after each Tixel or ResurFX treatment visit using the VAS questionnaire on a 0 to 10 scale
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tixel | Laser
Number analyzed (Participants) | 24 | 22
score on a scale
  tretament 1 | 4.6 (2.7) | 6.5 (2.1)
  treatment 2 | 4.2 (2.7) | 5.6 (2.8)
  treatment 3 | 4.2 (2.6) | 5.9 (2.6)
  treatment 4 | 3.2 (2.4) | 5.1 (2.0)
  treatment 5 | 2.9 (2.5) | 5.7 (2.0)

5. Secondary Outcome: Number on End-User Experience Scale
Description: The scores were converted to the same scale (a minimal score of 10 and a maximal score of 100 ) for both treatments, where a score of 10 is considered the wors outcome, and a score of 100 is considered the better outcome. For ResurFX, the maximal score is 45 therefore, the transformed score= total score *45 /100; for Tixel the maximal score is 50 therefore the transformed score =*50/100.
Time Frame: After performing 5 treatments with each device. After performing between 20 or 30 treatments with each device. After completing all the required treatments in the investigator's study site with both devices.
Population: End of user experience total score
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Tixel | Laser
Number analyzed (Participants) | 24 | 22
score on a scale
  After performing 5 treatments with each device. 100 excellent satisfaction. | 82.2 [10 to 100] | 62.0 [10 to 100]
  After performing between 20 or 30 treatments with each device. 100 excellent satisfaction. | 86.7 [10 to 100] | 80.0 [10 to 100]
  After completing all the required treatments in the investigator's study site with both devices. | 93.3 [10 to 100] | 93.0 [10 to 100]

6. Secondary Outcome: Mean Score Performance as Measured by the Fitzpatrick Classification of Facial Wrinkling (FWCS)
Description: The FWCS shall be assessed and quantified by the handling physician at study visits 1-8. The FWCS is classified as I-III, where I indicated mild/fine wrinkles and III indicates moderate wrinkles. (baseline to 42 weeks)
Time Frame: baseline, 42 Weeks
Population: Fitzpatrick Wrinkle Classification Score- Change
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tixel | Laser
Number analyzed (Participants) | 31 | 30
units on a scale | 0.5 (1.0) | 0.1 (0.9)

7. Secondary Outcome: Mean Improvement Performance as Measured by Improvement Global Assessment
Description: Improvement Global Assessment is scored on a scale from 1-4, with 1 indicating a poor response and 4 indicating an excellent response. This will be assessed at study visits 2-8. (from week 4- week 42)
Time Frame: visit 2, 3, 4, follow up 1, 2, 3
Population: global improvement assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tixel | Laser
Number analyzed (Participants) | 34 | 34
score on a scale
  treatment 2: number analyzed (Participants) | 31 | 30
  treatment 2 | 1.58 (0.62) | 1.6 (0.67)
  treatment 3: number analyzed (Participants) | 29 | 27
  treatment 3 | 1.86 (0.79) | 2.00 (0.83)
  treatment 4: number analyzed (Participants) | 17 | 17
  treatment 4 | 2.12 (0.78) | 2.29 (0.69)
  follow up 1: number analyzed (Participants) | 27 | 22
  follow up 1 | 1.89 (0.64) | 2.23 (0.87)
  follow up 2: number analyzed (Participants) | 23 | 15
  follow up 2 | 2.22 (0.82) | 2.47 (0.83)
  follow up 3: number analyzed (Participants) | 25 | 22
  follow up 3 | 2.20 (0.82) | 2.50 (1.01)

8. Secondary Outcome: Mean Score of Performance as Measured by 5-point Wrinkle Assessment Scale (WAS)
Description: The 5-point WAS is scored on a scale from 0-4, with 0 indicating no visible wrinkles and 4 indicating very deep wrinkles. This will be assessed at study visits 1-8. (baseline to 42 weeks)
Time Frame: 42 Weeks
Population: Skin assessments Changes from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tixel | Laser
Number analyzed (Participants) | 31 | 30
score on a scale | 0.3 (0.6) | 0.2 (0.4)

ADVERSE EVENTS:
Time Frame: 42 weeks
Arm/Group | Tixel | Laser
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 3/34 | 1/34
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tixel (N=34) | Laser (N=34)
Eye Dryness (Eye disorders) | 1 (1) | 0 (0) — Dry eye
Red eye (Eye disorders) | 1 (1) | 0 (0) — Ocular hyperemia
Watering eyes (Eye disorders) | 1 (1) | 0 (0) — Lacrimation increased
Uveitis (Eye disorders) | 0 (0) | 1 (1) — Uveitis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-24): https://cdn.clinicaltrials.gov/large-docs/72/NCT03454672/Prot_SAP_000.pdf